CLINICAL TRIAL: NCT06209931
Title: Retrograde Intrarenal Surgery With Tip Flexible Pressure-controlling Ureteral Access Sheath Versus Mini Percutaneous Nephrolithotomy for the Treatment of 2-3-cm Kidney Stones
Brief Title: RIRS With Tip Flexible Pressure-controlling Ureteral Access Sheath Versus Mini PCNLfor Kidney Stones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Ganzhou Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Huang Xin, Associate Senior Doctor, The Affiliated Ganzhou Hospital of Nanchang University
Other Study IDs: TY-ZKY-2023-045-12
Record Dates: First submitted 2023-12-09; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RIRS: Patients were performed under general anesthesia in the oblique supine lithotomy position. Initially, preliminary ureteroscopy was performed with a semirigid 8/9.8 Fr ureteroscope guided by zebra guide wire. Next, the patented tip flexible pressure-controlling ureteral access sheath (UAS,12/14 Fr) was inserted along the guidewire without the fluoroscopic guidance. The fully automatic mode was chosen to operate the platform.The pressure sensory and suctioning channels of UAS were connected to the irrigation and suctioning platform. After water injection, zero calibration was performed at platform. Perfusion flow rate was then set at 100-150 ml/min, the renal pelvic pressure (RPP) control value was set at -15~5 mmHg, the RPP warning value was set at 20 mmHg, and the RPP maximum value was set at 30 mmHg. Intraoperatively, a holmium laser was used to crush the stone at 1.5-2.0 J/pulse with a frequency of 20-30 pulses/s ( (CHUNHUI, CHINA, 276µm).
  Interventions: Procedure: RIRS
- MPCNL: Patients were performed under general anesthesia. The patient was first placed in a lithotomy position. A 5 Fr ureteral catheter was then inserted retrogradely into the renal pelvis through cystoscopy or ureteroscopy , and saline was continuously infused to produce artificial hydronephrosis. The patient was then placed in the prone position. Ultrasound-guided percutaneous punctures were made with an 18-gauge coaxial needle into the targeted calix. The puncture point was in the 12th rib infracostal margin, between the posterior axillary line and scapula line. A Zebra guidewire was inserted and fixed. The puncture needle was then removed. After a 0.5-0.7 cm skin incision was made, the percutaneous tract was dilated serially over the guidewire with a fascial dilator to 18Fr. Holmium laser lithotripsy at 1.5-2.0 J/pulse with a frequency of 20-30 pulses/s (CHUNHUI, CHINA, 550µm) was performed with a 18 Fr peel-away sheath.

INTERVENTIONS:
Procedure: RIRS — RIRS with tip flexible pressure-controlling ureteral access sheath versus mini PCNL for the treatment of 2-3-cm kidney stones
  Other Names: MPCNL
  Groups: RIRS

SUMMARY:
The goal of this observational study is to compare the safety and efficacy between RIRS with tip flexible pressure-controlling ureteral access sheath and mini percutaneous nephrolithotripsy（PCNL） for the treatment of 2-3-cm kidney stones.

DETAILED DESCRIPTION:
Retrograde Intrarenal Stone Surgery (RIRS) has become one of the most common treatments for renal stones. The development of ureteral access sheath (UAS) is a significant advance in RIRS. In recent years, various improvements have been made to UAS, especially the emergence of a suction UAS and a tip flexible UAS. Using the advantages of suction and tip flexible technology, our team developed a tip flexible pressure-controlling UAS, which significantly improves the safety and effectiveness of RIRS. However, the current guidelines can recommend the indication of RIRS in kidney stones less than 2cm, and percutaneous nephrolithotomy(PCNL) is still preferred for kidney stones larger than 2 cm. Therefore, this study is the first to compare the safety and efficacy between RIRS with tip flexible pressure-controlling UAS and mini PCNL in the treatment of 2 to 3 cm kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* American Society of Anesthesiology score 1-2
* Kidney stone diameter of 2-3 cm confirmed by CT
* Capable of giving written informed consent, which includes adherence with the requirements of the trial

Exclusion Criteria:

* Patients with abnormal urinary tract anatomy (such as horseshoe kidney or ileal conduit)
* Patients with uncontrolled UTI
* Patients with health or other factors that are absolute contraindications to RIRS or PCNL .Patients unable to understand or complete trial documentation.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney stones were confirmed in all patients by imaging, including urinary tract ultrasonography, intravenous urography, and computed tomography (CT). Stone size was calculated by CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Immediate stone-free rate | Postoperative day 1-7
  No residual stone or stone fragments less than 2 mm on low-dose CT scan at postoperative day 1-7 are defined as stone free.
Stone-free rate at 1 months | Postoperative 1 month
  No residual stone or stone fragments less than 2 mm on kidney, ureter, and bladder at 1 months are defined as stone free.
Complications up to 3 months post | Postoperative 3 month
Operation time | the time from the insertion of the suction sheath and renal puncture to the end of the operation,assessed up to 90 minutes.
  The operation time of RIRS and mini PCNL was defined as the time from the insertion of the suction sheath and renal puncture to the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Leming Song, Study Chair — The Affiliated Ganzhou Hospital of Nanchang University
Locations (1):
- Xiaolin Deng, Ganzhou, Jiangxi, China